CLINICAL TRIAL: NCT06816602
Title: The Effect of Structured Education Given to Individuals with Permanent Ostomy on Patient Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Özge İşeri (Other)
Responsible Party: Sponsor-Investigator, Özge İşeri, Assistant Professor, Ondokuz Mayıs University, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMU 2024/450; Ondokuz Mayıs University (Other: Ondokuz Mayıs University)
Record Dates: First submitted 2025-01-29; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Ostomy - Ileostomy or Colostomy
Keywords: ostomy; education; body image; sexual satisfaction; quality of life
MeSH Terms: conditions — Orgasm | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with single blinded experimental and control group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Control
- Experimental group (Experimental): Education
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: education — Receiving structured education
  Arms: Experimental group

SUMMARY:
Stoma is the surgical creation of an artificial opening on the abdominal surface for the purpose of evacuation. Although stomas are created to help individuals return to a healthy and productive life, to maintain a better quality and longer life and to improve the underlying pathology, they significantly affect the physical, mental, emotional and social life of patients. Stoma is also considered to be a very difficult situation to accept because it causes physical changes in individuals. Therefore, it causes problems in body image, sexual life and self-confidence that are difficult to cope with. In addition to these problems, changes in physical appearance and physiological problems as a result of stoma opening negatively affect the body image perception of the individual, cause him/her to see himself/herself different from others, feel ashamed of himself/herself, decrease self-esteem and self-confidence, feel fear of rejection by family and friends and limit social activities. Psychological disorders such as obsession, denial and imaginary rectum sensation are also seen in this period, and the patient may react with anger, anxiety, depression and isolation. In short, stoma negatively affects the quality of life and all physical, psychological, spiritual and social aspects of the individual. In a multicentre study, it was found that all aspects of quality of life of individuals had a decreasing score after stoma surgery. In a systematic review, it was shown that quality of life decreased after stoma formation for both cancer and non-cancerous reasons. Education and counselling interventions are very important for this. In a study, it was reported that telephone counselling had a positive effect on patients in order to prevent their concerns about sexual life and the difficulties they experienced with their stoma. However, there is no study in the literature that provides face-to-face structured training to individuals with permanent ostomy and monitors the effect of this training on body image, sexual satisfaction and quality of life. The aim of this study is to provide face-to-face structured education to patients with ostomy and to examine the effect of this education on body image, sexual satisfaction and quality of life.

DETAILED DESCRIPTION:
According to the data obtained from researches and associations in the USA, approximately 725,000-1,000,000 individuals are thought to have stoma today and this number is increasing day by day. In the United States, between 120,000-150,000 new stomas are opened every year. In Turkey, this number was reported to be 2509 individuals in the statistics made in 2017. Although stoma is applied to prolong the life span of patients, to help them return to the living standards they had before diagnosis, to improve their quality of life and to improve the underlying pathology, it causes them to encounter problems that cause changes in lifestyle in physical, emotional, sexual, psychological and social aspects. Studies have shown that the quality of life of individuals after stoma surgery has a decreasing score in all aspects and in another study, it was reported that telephone counselling had a positive effect on patients to prevent their concerns about sexual life and the difficulties they experienced with their stoma. The uniqueness of this study is that face-to-face structured training was given to patients with permanent ostomy and the effect on body image, sexual satisfaction and quality of life of individuals in the first and third months was examined.

ELIGIBILITY:
Inclusion Criteria: Over 18 years old, with a permanent ostomy, with ileostomy or colostomy, no cognitive or mental problems Exclusion Criteria: Previous structured training on living with a stoma, those with psychiatric or mental problems, those undergoing revision surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
body image | pretest, 1 month after intervention, 3 month after intervention
  Body Image Scale; It was developed by Hopwood (2001) and adapted to Turkish by Karayurt et al. (2015). The scale consists of 10 questions that question patients' perceptions of their individual body image and their reactions to change. A low scale score indicates that the perception of self-image is better. Cronbach Alpha value in the Turkish version of the scale is 0.94. Item-Total Score Correlation Coefficients vary between 0.75 and 0.91.
Sexual Satisfaction | pretest, 1 month after intervention, 3 month after intervention
  Golombuk-Rust Sexual Satisfaction Scale: Golombuk-Rust (Rust and Golombok 1986) sexual satisfaction scale is a scale used to evaluate sexual problems and their severity consisting of 28 questions. It consists of 12 sub-assessment scales related to empotence, premature ejaculation, orgasm disorder, vaginismus, miscommunication, frequency and male and female avoidance, male and female insensitivity and male and female dissatisfaction. Scores of five and above indicate impairment in sexual functions in that sub-dimension. Tuğrul et al. (1993) reported that the Golombuk-Rust Sexual Satisfaction Scale is valid and reliable in our country.
Quality of Life | pretest, 1 month after intervention, 3 month after intervention
  Quality of Life Scale for Individuals with Ostomy (QoLQS): It was developed by Baxter et al. (2006). The scale, which evaluates the quality of life of individuals with stoma, was translated into Turkish by Karadağ et al. in 2011. It was found that the Stoma Quality of Life Scale, which consisted of a total of 19 items and 3 subscales, was valid and reliable for adult individuals with stoma (ileostomy, colostomy and urostomy) in the Turkish population. The reliability coefficient of the scale (Cronbach α) was found to be 0.87 and the reliability coefficients of the subscales were 0.77, 0.72 and 0.76, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs Unıversity, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No